CLINICAL TRIAL: NCT06646367
Title: Effect of Alexander Technique on Neck Pain and Quality of Life in Lactating Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aml Elsaid Hamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005325
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): It will include 36 lactating females suffering from neck pain who will receive conventional therapy in the form of moist heat for 30 min, 5 times per week for 5 weeks and transcutaneous electrical nerve stimulation (TENS) that will be applied for 25 min, 5 times per week for 5 weeks.
  Interventions: Other: Conventional therapy
- Conventional therapy + Alexander technique (Experimental): It will include 36 lactating females suffering from neck pain who will receive the same conventional therapy in addition to the Alexander technique which will be applied for 60 min, 2 classes per week, for 5 weeks.
  Interventions: Other: Conventional therapy; Other: Alexander technique

INTERVENTIONS:
Other: Conventional therapy — All participants in the two groups will receive conventional therapy in the form of TENS and moist heat for 5 weeks.TENS will be applied 5 times a week for 5 weeks at a frequency of 80Hz with 10- to 30-mA intensity for 25 minutes. Four surface electrodes (5x5 cm each) were situated over the painful region in the neck (two electrodes will be placed in either side of the spine high on neck, just underneath the skull and the other two electrodes will be placed about 5cm underneath them) with intensity in the tactile sensation threshold. The hot packs will be applied for 30 minutes on the cervical area, 5 times per week for 5 weeks.
Other: Alexander technique — Women in the experimental group will attend 10 Alexander Technique classes (60 minutes each, twice a week for 5 weeks). The Alexander Technique focuses on body awareness, reducing muscle tension, and improving coordination through three principles: enhanced awareness, purposeful inhibition, and mental imagery. Participants will learn to release habitual muscle tension and explore alternative movement patterns, covering biomechanics and ergonomics of the neck, spine, and limbs. The sessions involve hands-on guidance, verbal instruction, and group activities. Daily practice in a semi-supine position is encouraged to improve posture, coordination, and overall well-being.
  Arms: Conventional therapy + Alexander technique

SUMMARY:
This study will be conducted to investigate the effect of the Alexander technique on neck pain and quality of life in lactating women.

DETAILED DESCRIPTION:
During breastfeeding, incorrect positioning and placement of hands to support the baby's weight can irritate the musculature of the hands. Repeating the same position frequently can lead to radiating pain in the elbows and hands. Additionally, adopting different postures to compensate for the pain while sitting, standing, or lying down can cause mechanical changes in the cervical, thoracic, and lumbar spine, altering the body's correct posture.

The Alexander Technique is a non-exercise approach focused on improving the modulation of postural muscle activity. It offers an individualized approach to developing skills that help people recognize, understand, and avoid poor habits that affect postural tone and neuromuscular coordination. Its lessons are associated with clinically relevant long-term reductions in neck pain and disability.

Some previous studies examined effect of Alexander technique on neck pain and on quality of life in different population, but in our knowledge this is the first study will be conducted to investigate effect of Alexander technique on neck pain and quality of life in lactating women, so this study will be conducted to provide an insight about the beneficial effect of the Alexander Technique on neck pain and quality of life in lactating women which will be of valuable benefits in the women's health field.

ELIGIBILITY:
Inclusion Criteria:

* Lactating females experiencing neck pain (six weeks to 1year postpartum).
* Able to understand and follow the Alexander Technique instructions.
* Their age will be ranged from 20-35 years old.
* Their BMI will be less than 30 kg/m2 .
* Their pain level is ≥ 4 on numeric pain rating scale.
* They have mild disability on Neck Disability Index Questionnaire (NDI).
* They have limited cervical range of motion (the normal flexion range of motion is 80° to 90°, extension 70°, lateral flexion 20° to 45°, and rotation up to 90°).

Exclusion Criteria:

* Neck pain as consequence of disc protrusion or prolapse, whiplash, congenital deformity of the spine, spinal stenosis, neoplasm, inflammatory rheumatic disease, neurological disorder, and psychosis.
* Women who had invasive treatment of the spine within the previous three weeks, or spinal surgery or presence of neck history of trauma.
* Presence of contraindications to spinal movement, such as fracture or dislocation.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of neck pain intensity | 5 weeks
  The pain intensity will be assessed through numeric pain rating scale for all participating women in both groups before and after the treatment program. The woman will be asked to circle the number between 0 (represents no pain) and 10 (represents the worst pain) that best represents their pain intensity. She will be asked to indicate the intensity of her current, best, and worst pain levels over the past 24 hours on the scale, the mean of these three ratings is calculated to represent the patient's overall pain intensity.
Quality Of Life assessment | 5 weeks
  The Short Form Survey Instrument (SF-36) will be used to assess the health-related quality of life for all women in both groups before and after the treatment program. The SF-36 is a self-administered questionnaire containing 36 items, which takes about five minutes to complete. It measures health across eight multi-item dimensions, covering functional status, well-being, and overall health evaluation, each associated with 2-10 possible answers. The response to each question is extrapolated to a standardized set of answers, and the results are transferred to a scale of 0-100, where 0 represents the worst state of health and 100 represents the best state of health measured. It has good validity and reliability and can be used as a general questionnaire to assess quality of life.

SECONDARY OUTCOMES:
Measurement of neck flexion range of motion (ROM) | 5 weeks
  The goniometer will be used to measure flexion ROM for all women in both groups before and after the treatment program. Ask the patient to sit up straight in a chair with their feet flat on the floor, their arms hanging down by their sides, and their thoracic spine resting against the back of the chair. Place the goniometer's axis over the external auditory meatus before using it. Place the stationary arm perpendicular to the floor or vertically. Place the movable arm in line with the nose's base. This should be noted as 0°. For measuring cervical flexion ROM ask the woman to nod forward and lift their chin up to their chest,
Measurement of neck extension range of motion (ROM) | 5 weeks
  The goniometer will be used to measure extension ROM for all women in both groups before and after the treatment program. Ask the patient to sit up straight in a chair with their feet flat on the floor, their arms hanging down by their sides, and their thoracic spine resting against the back of the chair. Place the goniometer's axis over the external auditory meatus before using it. Place the stationary arm perpendicular to the floor or vertically. Place the movable arm in line with the nose's base. This should be noted as 0°. For measuring cervical extension ROM ask the woman to stare as far upward as she can until her neck is fully extended.
Measurement of neck lateral flexion range of motion (ROM) | 5 weeks
  The goniometer will be used to measure lateral flexion ROM for all women in both groups before and after the treatment program. The goniometer fulcrum will be aligned over the spinous process of the C7. The fixed arm of the goniometer will be aligned vertically along the imaginary line between the two acromion processes. The movable arm will be aligned over the external occipital protuberance. Then, instruct the woman to flex his/her neck laterally and record readings of the goniometer at each extreme of the motion in both sides.
Measurement of neck rotation range of motion (ROM) | 5 weeks
  The goniometer will be used to measure rotation ROM for all women in both groups before and after the treatment program. The goniometer fulcrum will be aligned over the center of the subject's head, the fixed arm of the goniometer will be aligned with an imaginary line between the subject's acromion processes and the movable arm will be aligned with the tip of the subject's nose. The woman will be told to stare directly her head, ideally at eye level. Next, instruct the woman to turn her head as far to the left as she can without tipping or tilting it. Take goniometer readings at both ends of the motion and record them and repeat the procedure for the opposite direction.
Assessment of neck function | 5 weeks
  Neck Disability Index (NDI) will be used for all women in both groups before and after treatment program to assess self-rated disability, including aspects beyond current pain levels, by evaluating an individual's ability to perform daily activities. Each woman will be asked to choose from NDI questionnaire which comprises 10 items, each scored on a scale of 0 to 5, resulting in a maximum total score of 50. Lower scores reflect less self-rated disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohamed Hanfy, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt